CLINICAL TRIAL: NCT07134751
Title: Febrile Infants Swedish Study
Acronym: FISS
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Orfanos Ioannis, MD, PhD, Senior Consultant Pediatrician, Region Skane
Other Study IDs: Dnr 2024-05132-02
Record Dates: First submitted 2025-08-05; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Febrile Illness Acute; Meningitis, Bacterial; Urinary Tract Infection (Diagnosis); Invasive Bacterial Infection; Serious Bacterial Infection; Bacteremia; Sepsis
Keywords: Guidelines; Febrile infants; Age ≤60 days; Management; Serious Bacterial Infections; Invansive Bacterial Infections; Clinical prediction tool
MeSH Terms: conditions — Meningitis, Bacterial; Urinary Tract Infections; Disease; Bacteremia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Febrile Infants aged ≤60 days: Febrile Infants aged ≤60 days who present to the pediatric emergency department

SUMMARY:
Approximately one million febrile infants aged ≤60 days present annually to pediatric emergency departments (PEDs) in Europe and the United States. Although fewer than 5% are diagnosed with meningitis or bacteremia (invasive bacterial infections - IBIs), and 10-15% with urinary tract infections (UTIs), current guidelines recommend extensive diagnostic evaluations, hospitalization, and empirical treatment with broad-spectrum parenteral antibiotics. This approach may contribute to medical overuse, with implications for patient care, healthcare resource utilization, and environmental sustainability.

The Febrile Infants Swedish Study (FISS) is a prospective observational study conducted across 11 PEDs in Sweden. All febrile infants aged ≤60 days presenting to participating sites will be eligible. A new clinical guideline for the management of infants with fever without source (FWS) will be implemented in 7 PEDs, while 4 PEDs will continue with current standard practice and serve as a comparison group.

The study is expected to run for approximately two years and aims to recruit a minimum of 2,500 febrile infants

DETAILED DESCRIPTION:
BACKGROUND

Each year, around one million febrile infants aged ≤60 days present to pediatric emergency departments (PEDs) in Europe and the United States. Previous studies report that 2-5% of these infants are diagnosed with meningitis or bacteremia (invasive bacterial infections - IBIs) and 10-15% with urinary tract infections (UTIs). Due to the potential severity of these infections, current guidelines recommend comprehensive diagnostic evaluations, hospitalization, and empirical treatment with broad-spectrum antibiotics. Consequently, an estimated 800,000 infants undergo these interventions annually without confirmed SBI.

These practices may have unintended consequences. Lumbar punctures can be painful, stressful, and time-consuming, with unsuccessful attempts linked to longer hospital stays. Early antibiotic exposure has been associated with increased risks of chronic conditions and reduced vaccine response and contributes to antimicrobial resistance. Hospitalization may lead to complications, disrupt breastfeeding, and impose financial and emotional burdens on families. Routine testing can result in overdiagnosis and medical overuse. Additionally, healthcare delivery has environmental implications, with each hospital bed-day generating significant waste and energy consumption.

Current guidelines rely on binary thresholds for biomarkers such as CRP and procalcitonin. They also lack consideration of clinical context, such as the infant's condition or fever characteristics, resulting in a uniform approach that may not suit individual cases.

There is a need for more individualized, evidence-based guidelines that integrate clinical and laboratory findings to support risk stratification and informed decision-making. Guidelines that reduce unnecessary interventions may improve care, optimize resource use, and lessen environmental impact.

The Febrile Infants Swedish Study (FISS) aims to evaluate a new clinical guideline.

PRIMARY AIM

To evaluate the new guideline for the management of infants aged ≤60 days and compare to current praxis.

SECONDARY AIMS

* To collect clinical data (height/duration of fever, gestational age, birth weight, clinical symptoms/signs, laboratory results, diagnoses) which will enable the improvement of the guideline and the development of a more individualized management guideline.
* To describe adherence to the new guideline and variation between the study sites in the management of febrile infants aged ≤60 days.

STUDY DESIGN

This will be a multicenter prospective observational study in 11 PEDs in Sweden. All febrile infants presented to the study PEDs will be considered as eligible for the study. The new guideline will be implemented as the PEDs standard management protocol for infants aged ≤60 days with FWS in 7 PEDs (Lund, Malmö, Helsingborg, Kristianstad, Ystad, Örebro, Sachsska-Stockholm). In 4 PEDs (Uppsala, Gothenburg, Jönköping, and Karolinska-Stockholm), the management of febrile infants aged ≤60 days will continue according to current praxis and these PEDs will participate in this study as a control group

STUDY POPULATION

All febrile infants aged ≤60 days brought to any of the study PEDs will be considered eligible for the study.

INCLUSION CRITERIA

1. Age ≤60 days.
2. Temperature ≥38.0 C measured either at home or at the PED.

DEFINITIONS

Fever Without a Source (FWS): Defined as a body temperature ≥38°C, measured either at home or in the pediatric emergency department (PED), without an identifiable focus of infection following medical history and physical examination.

Serious bacterial infection (SBI) is defined as a Urinary Tract Infection (UTI), bacteremia, or bacterial meningitis.

Urinary tract infection (UTI) is defined as urine dipstick positive for leukocyte esterase or nitrite and a urine culture with growth of (1) any amount of a single pathogen in samples obtained by suprapubic aspiration; (2) ≥10,000 colony- forming units (cfu)/ml of a single pathogen in samples obtained by a 'clean catch' method or catheterization.

Bacteremia is defined as growth of a bacterial pathogen in a blood culture. The presence of coagulase- negative staphylococci, Propionibacterium spp, Bacillus cereus spp, micrococci, alpha haemolytic streptococci and diphtheroids were considered contaminants, unless indicated otherwise because of clinical or laboratory parameters.

Bacterial meningitis is defined by the presence of a cerebrospinal fluid (CSF) culture or a CSF polymerase chain reaction (PCR) test positive for a bacterial pathogen. Cases with indirect clinical or laboratory indications of bacterial meningitis, such as elevated CSF cell count with positive blood culture and negative CSF culture/PCR, especially if antibiotics are given before the lumbar puncture, can be considered as bacterial meningitis,

Invasive bacterial infection (IBI) is defined as bacterial meningitis or bacteremia.

Delayed treated SBI will be regarded in infants with an SBI who did not receive broad-spectrum antibiotics at the initial management.

ELIGIBILITY:
Inclusion Criteria:

* Temperature ≥38.0 C (measured either at home or at the pediatric emergency department)
* Age ≤60 days

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All febrile infants aged ≤60 days brought to any of the study Pediatric Emergency Departments will be considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of febrile infants aged ≤60 days with meningitis, bacteremia, and urinary tract infection identified by the new guideline and the proportion of those that received treatment with delay. | 10 days of attendance

SECONDARY OUTCOMES:
The proportion of investigations, antibiotic treatments, and hospitalizations among febrile infants aged ≤60 days who visited the PED. | Day 1
The prevalence of meningitis, bacteremia, and urinary tract infection among febrile infants aged ≤60 days. | 10 days of attendance
Duration and height of the fever, gestational age, birth weight, breastfeeding, clinical signs and symptoms, and laboratory results. | Day 1

CONTACTS AND LOCATIONS:
Locations (11):
- Sweden (11):
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Ryhov County Hospital, Jönköping
  - Kristianstad Central Hospital, Kristianstad
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Sachs' Children and Youth Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
  - Ystad Hospital, Ystad

IPD SHARING:
Plan to Share IPD: Yes
Anonymised datasets not containing any personal data will be available after publication upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 2 years and ending 4 years after the publication of results